CLINICAL TRIAL: NCT07316751
Title: Italian Translation and Validation of the GIDS-PD Scale for Parkinson's Disease
Acronym: GIDS-PD_ITA
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: GIDS-PD_ITA
Record Dates: First submitted 2025-11-24; First posted 2026-01-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: PARKINSON DISEASE (Disorder); Parkinson Disease
Keywords: Parkinson's Disease; Gastrointestinal Dysfunction; Scale Validation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to translate and validate the Gastrointestinal Dysfunction Scale for Parkinson's Disease (GIDS-PD) into Italian to enable the assessment of gastrointestinal symptoms in Italian-speaking patients with Parkinson's disease. The psychometric properties of the translated instrument will be evaluated through a multi-phase process involving translation/back-translation, pre-testing, and large-scale validation across multiple Italian centers

DETAILED DESCRIPTION:
Gastrointestinal dysfunction is a frequent and burdensome non-motor feature of Parkinson's disease, yet validated tools to measure these symptoms are not available for Italian-speaking patients. The study will will undergo three distinct phases, as specified by the MDS guidelines (International Parkinson and Movement Disorder Society, 2023): translation and back-translation (Phase I), pre-test (Phase II), large-scale validation test (Phase III).

* Phase I The translation and back-translation process will be conducted by two independent teams; one team will translate the content from English to Italian, followed by another team independently back-translating it from Italian to English (back-translation).
* Phase II Phase II will involve about 10 PD patients, as heterogeneous as possible, from different Italian regions, and 10 clinicians (PD nurses, neurologists, etc) examiners. The instrument, in this preliminary version, will be presented to a group of about 10 PD patients for the pre-test phase. This phase will be used to establish the basic psychometric properties of the scale and identify items that could potentially be culturally complex.
* Phase III Once the official translation has been approved, the instrument will be administered to a sample of PD patients, native Italian speakers, heterogeneous as far as possible in age and gender.

The final Italian version will be assessed for data quality, acceptability, construct validity, and reliability in a cohort of patients diagnosed with Parkinson's disease across multiple Italian centers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of PD according to the Movement Disorder Society (MDS) diagnostic criteria (Postuma RB et al., 2015);
* Italian-native patients or patients that understand Italian correctly at least;
* Participants mentally and physically able to understand and sign the informed consent form.

Exclusion Criteria:

* Persons in the terminal phase of disease;
* Persons with clinically relevant cognitive impairment;
* Persons diagnosed with Parkinsonism other than PD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients with PD attending the movement disorders Units of the study centres.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Translation the Italian version of GIDS-PD | 3 years
  Score on the Italian version of the Geriatric Impulse Dyscontrol Scale-Parkinson's Disease (GIDS-PD), total score ranging from 0 to 100, with higher scores indicating greater impulse control difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Eleopra, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (5):
- Italy (5):
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Ospedale Universitario Luigi Sacco, Milano, Italia, Milan
  - Unità Parkinson e Disturbi del Movimento, Dipartimento di Neuroscienze(DNS), Università di Padova, Padova, Italia, Padua
  - Centro per le Malattie Neurodegenerative e l'Invecchiamento Cerebrale, Università degli Studi di Bari "Aldo Moro" presso la Pia Fondazione "Card. G. Panico", Tricase, Italia, Tricase
  - Unità di Neurologia, Divisione Malattia di Parkinson e Disturbi del Movimento, Dipartimento di Neuroscienze, Biomedicina e Scienze del Movimento, Università di Verona, Italia, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Leta V, Klingelhoefer L, Longardner K, Campagnolo M, Levent HC, Aureli F, Metta V, Bhidayasiri R, Chung-Faye G, Falup-Pecurariu C, Stocchi F, Jenner P, Warnecke T, Ray Chaudhuri K; International Parkinson and Movement Disorders Society Non-Motor Parkinson's Disease Study Group. Gastrointestinal barriers to levodopa transport and absorption in Parkinson's disease. Eur J Neurol. 2023 May;30(5):1465-1480. doi: 10.1111/ene.15734. Epub 2023 Mar 7. PMID 36757008
- [Background] Metta V, Leta V, Mrudula KR, Prashanth LK, Goyal V, Borgohain R, Chung-Faye G, Chaudhuri KR. Gastrointestinal dysfunction in Parkinson's disease: molecular pathology and implications of gut microbiome, probiotics, and fecal microbiota transplantation. J Neurol. 2022 Mar;269(3):1154-1163. doi: 10.1007/s00415-021-10567-w. Epub 2021 Apr 21. PMID 33881598
- [Background] Maxwell SE, Kelley K, Rausch JR. Sample size planning for statistical power and accuracy in parameter estimation. Annu Rev Psychol. 2008;59:537-63. doi: 10.1146/annurev.psych.59.103006.093735. PMID 17937603
- [Background] Camacho M, Greenland JC, Williams-Gray CH. The Gastrointestinal Dysfunction Scale for Parkinson's Disease. Mov Disord. 2021 Oct;36(10):2358-2366. doi: 10.1002/mds.28675. Epub 2021 Jun 16. PMID 34133059
- [Background] Bhidayasiri R, Phuenpathom W, Tan AH, Leta V, Phumphid S, Chaudhuri KR, Pal PK. Management of dysphagia and gastroparesis in Parkinson's disease in real-world clinical practice - Balancing pharmacological and non-pharmacological approaches. Front Aging Neurosci. 2022 Aug 11;14:979826. doi: 10.3389/fnagi.2022.979826. eCollection 2022. PMID 36034128